CLINICAL TRIAL: NCT02506777
Title: Phase II Multicenter Randomized Study to Compare Neoadjuvant FDC With Melatonin or Metformin Versus FDC Alone in The Therapy of Locally Advanced Breast Cancer.
Brief Title: Neoadjuvant FDC With Melatonin or Metformin for Locally Advanced Breast Cancer.
Acronym: MBC1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBC1
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Melatonin, metformin, chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Fluorouracil; Doxorubicin; Cyclophosphamide; Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FDC x 6 cycles with metformin (Experimental): 32 patients will receive 5 - Fluoruracil 500 mg/m^2, doxorubicin 50 mg/m^2, cyclophosphamide 500 mg/m^2 once every 21 days with metformin 850 mg BID
  Interventions: Drug: metformin; Drug: Fluoruracil; Drug: Doxorubicin; Drug: Cyclophosphamide
- FDC x 6 cycles with melatonin (Experimental): 32 patients will receive 5 - Fluoruracil 500 mg/m^2, doxorubicin 50 mg/m^2, cyclophosphamide 500 mg/m^2 once every 21 days with melatonin 3 mg before sleep daily
  Interventions: Drug: Fluoruracil; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: melatonin
- FDC x 6 cycles (Active Comparator): 32 patients will receive 5 - Fluoruracil 500 mg/m^2, doxorubicin 50 mg/m^2, cyclophosphamide 500 mg/m^2 once every 21 days
  Interventions: Drug: Fluoruracil; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: metformin
  Other Names: siofor 850
  Arms: FDC x 6 cycles with metformin
Drug: Fluoruracil
Drug: Doxorubicin
  Other Names: Adriablastin
Drug: Cyclophosphamide
  Other Names: endoxan
Drug: melatonin
  Other Names: melaxen
  Arms: FDC x 6 cycles with melatonin

SUMMARY:
This study evaluates the addition melatonin and metformin to conventional chemotherapy FDC (Fluoruracil, Doxorubicin, cyclophosphamide) in the treatment of locally advanced breast cancer. Third of patients will receive FDCх6 cycles, other third will receive combination of melatonin and FDCх6 cycles and other patients will receive combination of metformin and FDCх6 cycles.

DETAILED DESCRIPTION:
The treatment of locally advanced breast cancer is a complicated issue. For neoadjuvant treatment is often needed to downstage locally advanced BC tumors prior to surgery, however many patients do not achieved objective response during treatment. The ability of melatonin and metformin to decrease side effects of chemotherapy had been investigated, moreover several studies confirm, that this drugs in combination with conventional treatment may increase objective response. But, this data is still controversial. We hypothesized that combinations of melatonin and conventional chemotherapy regimen such as FDC could be more effective than FDC alone in terms of response rate.

ELIGIBILITY:
Inclusion Criteria:

* Age >18. Obtained Inform Consent Morphologically confirmed breast cancer stage IIB, IIIA,IIIB,IIIC. ( triple negative, luminal B) Eastern Collaborative Oncology Group Performance Status Scale 0 - 2. Expected survival >6 month Adequate liver and bone marrow function

Exclusion Criteria:

* Systemic treatment for breast cancer IV stage disease Evidence of liver and bone marrow clinically meaningful disfunction Severe uncontrolled concomitant conditions and diseases Pregnancy or lactation Second malignancy Diabetes mellitus requiring drug therapy Any condition preventing study participation by investigator opinion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 months after FPFV
  Response will evaluate by RECIST criteria
Pathomorphological response | 6 months after FPFV
  Pathomorphological response will assess after surgery by Miller and Payne Scale

SECONDARY OUTCOMES:
Adverse events incidence | Until 30 days after last patient treatment visit
  Incidence of AE classified using NCI Common Terminology Criteria for AE v4

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir F Semiglazov, MD, PhD, DSc, Professor, Study Director — N.N. Petrov Research Institute of Oncology; Tatiana Y Semiglazova, Principal Investigator — N.N. Petrov Research Institute of Oncology
Locations (1):
- N.N. Petrov Research Institute of Oncology Clinical Diagnostic Department, Saint Petersburg, Russia